CLINICAL TRIAL: NCT02491580
Title: Post-transplant Cancer Incidence and Survival in Patients With or Without Pre-transplant Cancer
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: PreTXCa
Record Dates: First submitted 2015-06-30; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Neoplasms; Kidney Failure
MeSH Terms: conditions — Neoplasms; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- KTx Uppsala: Patients who have received a kidney transplant in Uppsala.
- KTx Europe: Patients who have received a kidney transplant in Uppsala.

SUMMARY:
Patients with previous malignancies have increasingly been accepted for renal transplantation. However, post-transplant malignancy risk and survival rates of these patients are unknown. Our aim was to assess if previous malignancies pose an unnecessarily high risk of post-transplant malignant tumours and if the organs as a resource are too limited for investment in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplanted patients from January 1982 through December 2013 with or without a pre transplant cancer.

Exclusion Criteria:

* Simultaneous kidney+pancreas transplantation.
* Islet cell transplanted patients
* Undiagnosed malignancies at the time of transplantation
* Death within a week after transplantation
* First transplantation at another hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplanted patients in Uppsala or Europe with or without a pre-transplant cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2370 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence of post-transplant cancer | Up to 33 years starting in January 1982.

SECONDARY OUTCOMES:
Patient survival | Up to 33 years starting in January 1982.
Cancer-induced mortality | Up to 33 years starting in January 1982.

OTHER OUTCOMES:
Graft survival | Up to 33 years starting in January 1982.

CONTACTS AND LOCATIONS:
Overall Officials: Vivan Hellström, MD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Department of Surgical Sciences, Section of Transplantation Surgery, Uppsala, Sweden

REFERENCES:
- [Derived] Hellstrom V, Lorant T, Dohler B, Tufveson G, Enblad G. High Posttransplant Cancer Incidence in Renal Transplanted Patients With Pretransplant Cancer. Transplantation. 2017 Jun;101(6):1295-1302. doi: 10.1097/TP.0000000000001225. PMID 27163539